CLINICAL TRIAL: NCT04839263
Title: Fast-track in Minimally Invasive Gynaecology: a Randomized Trial Comparing Costs and Clinical Outcomes
Brief Title: Fast-track in Minimally Invasive Gynaecology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Shahzia Lambat, Chief resident, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCER 15-103
Record Dates: First submitted 2021-03-31; First posted 2021-04-09 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Gynecologic Disease
Keywords: fast-track; laparoscopic hysterectomy; hospital costs
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Intervention Model Description: "FAST TRACK" protocol Preoperative evaluation and information
  Patient general health state optimization proposal prior to hospitalization:
  Preoperative strategy:
  * Hospitalization on surgery day
  * No prolonged fasting
  Perioperative strategy:
  * Pain control based on limited systemic opioid therapy use
  * Anti-nausea prophylaxis
  * Anaesthesia via IV propofol / remifentanyl
  * Bladder catheter removal postoperative
  Postoperative strategy:
  * Pain control using balanced analgesia
  * Gum chewing
  * Early oral refeeding and rapid mobilization
  * Venflon removal 6 hours post-op 2) "Conventional setting" protocol
  Preoperative strategy:
  * Hospitalization on surgery day
  * Fasting as of midnight prior to the day of surgery
  Perioperative strategy:
  - Balanced anaesthesia via halogens gases
  Postoperative strategy:
  * Same day refeeding and mobilization minimum 6 hours post operation
  * Bladder catheter and Venflon removal on day 1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "FAST TRACK" protocol (Active Comparator): "FAST TRACK" protocol Preoperative evaluation and information
  Patient general health state optimization proposal prior to hospitalization:
  Preoperative strategy:
  * Hospitalization on surgery day
  * No prolonged fasting
  Perioperative strategy:
  * Pain control based on limited systemic opioid therapy use
  * Anti-nausea prophylaxis
  * Anaesthesia via IV propofol / remifentanyl
  * Bladder catheter removal postoperative
  Postoperative strategy:
  * Pain control using balanced analgesia
  * Gum chewing
  * Early oral refeeding and rapid mobilization
  * Venflon removal 6 hours post-op
  Interventions: Procedure: "FAST TRACK" protocol
- "Conventional setting" protocol (No Intervention): "Conventional setting" protocol
  Preoperative strategy:
  * Hospitalization on surgery day
  * Fasting as of midnight prior to the day of surgery
  Perioperative strategy:
  - Balanced anaesthesia via halogens gases
  Postoperative strategy:
  * Same day refeeding and mobilization minimum 6 hours post operation
  * Bladder catheter and Venflon removal on day 1

INTERVENTIONS:
Procedure: "FAST TRACK" protocol — Preoperative evaluation and information
  Patient general health state optimization proposal prior to hospitalization:
  Preoperative strategy:
  * Hospitalization on surgery day
  * No prolonged fasting
  Perioperative strategy:
  * Pain control based on limited systemic opioid therapy use
  * Anti-nausea prophylaxis
  * Anaesthesia via IV propofol / remifentanyl
  * Bladder catheter removal postoperative
  Postoperative strategy:
  * Pain control using balanced analgesia
  * Gum chewing
  * Early oral refeeding and rapid mobilization
  * Venflon removal 6 hours post-op
  Arms: "FAST TRACK" protocol

SUMMARY:
Objective: Evaluate the effects of a fast-track (FT) protocol on costs and postoperative recovery.

Design: randomized trial

Setting: University Hospitals

Population: 170 women undergoing total laparoscopic hysterectomy for a benign indication

Methods: A FT protocol included the combination of minimally invasive surgery, analgesia optimization, early oral refeeding and rapid mobilization of patients was compared to a usual care protocol.

Main outcomes measure: Primary outcome was costs. Secondary outcomes were length of stay, postoperative morbidity and patient satisfaction.

DETAILED DESCRIPTION:
1. Fast-Track protocol:

   Preoperative
   * Anesthetic consultation
   * Proposal of optimization of patient's general health state + family meeting if necessary
   * Hospitalization on day of surgery
   * Solids stopped 6 hours prior to surgery, drinking encouraged up to 2 hours prior to surgery

   During surgery
   * Anti-infectious prophylaxis
   * Anesthesia via IV propofol/remifentanil
   * Anti-nausea prophylaxis
   * Pain control based on limited systemic opioid use

   Postoperative
   * Balanced analgesia for pain control
   * Antithrombotic prophylaxis
   * Early oral refeeding
   * Rapid mobilization
   * Gum chewing
   * Foley catheter removal at the end of surgery
   * Peripheral IV catheter removal 6 hours postoperatively
2. Usual care protocol :

Preoperative

* Anesthetic consultation
* Hospitalization on day of surgery
* Fasting beginning at midnight prior to surgery

During surgery

* Anti-infectious prophylaxis
* Balanced anesthesia via halogen gas
* Anti-nausea medication if needed

Postoperative

* Balanced analgesia for pain control
* Antithrombotic prophylaxis
* Same-day refeeding according to patient's wish
* Same-day mobilization according to patient's wish
* Foley and peripheral IV catheter removal on day 1 postoperatively

ELIGIBILITY:
Inclusion Criteria:

* women undergoing total laparoscopic hysterectomy for a benign indication

Exclusion Criteria:

* the requirement for an additional surgical procedure, such as prolapse repair or urinary incontinence, because a prolonged operative time could compromise early patient discharge and
* the inability to speak French because the patients were required to complete their data collection logbook in French.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women undergoing total laparoscopic hysterectomy for a benign indication
Enrollment: 170 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Hospital costs and ambulatory costs | Up to 1 month postoperative
  The economic evaluation covered hospital inpatient surgical care costs and ambulatory costs. Resource inputs were divided into two main categories: (1) hospital inpatient surgical costs and (2) ambulatory costs further divided into (2a) hospital-related costs (A&E Department consultations and hospital readmission) and (2b) community costs (community health + social costs and caregiver's loss of production costs). Hospital costs were collected using a computerized hospital information system developed by the University Hospitals of Geneva. The patients recorded community costs in a logbook containing the community health and social invoices and caregivers' number of absent working days. Caregivers' loss of production was extrapolated via Switzerland's median wage per working day.

SECONDARY OUTCOMES:
Hospital length of stay | Up to 1 month postoperative
  Hospital stay was retrieved from the computerized patient record
Postoperative morbidity rate during the first postoperative month | Up to 1 month postoperative
  Morbidity during the first postoperative month was monitored via patient consultations at the Accident and Emergency (A&E) Department
Satisfaction assessed by a three-point likert scale | Up to 1 month postoperative
  Patient satisfaction was evaluated on their day of discharge and at their 1-month postoperative follow-up visit based on a three-point likert scale regarding their satisfaction with the care they received. The likert scale ranged from 0 (unsatisfied) to 2 (satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Shahzia Lambat, Principal Investigator — HUG
Locations (2):
- Switzerland (2):
  - HUG, Geneva
  - University Hospitals, Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Bardram L, Funch-Jensen P, Jensen P, Crawford ME, Kehlet H. Recovery after laparoscopic colonic surgery with epidural analgesia, and early oral nutrition and mobilisation. Lancet. 1995 Mar 25;345(8952):763-4. 2. Basse L, Hjort Jakobsen D, Billesbølle P, Werner M, Kehlet H. A clinical pathway to accelerate recovery after colonic resection. Ann Surg. 2000 Jul;232(1):51-7. 3. Kehlet H, Wilmore DW. Multimodal strategies to improve surgical outcome. Am J Surg. 2002 Jun;183(6):630-41. 4. Kehlet H, Büchler MW, Beart RW Jr, Billingham RP, Williamson R. Care after colonic operation--is it evidence-based? Results from a multinational survey in Europe and the United States. J Am Coll Surg. 2006 Jan;202(1):45-54. 5. Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, et al. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77.
- [Derived] Lambat Emery S, Brossard P, Petignat P, Boulvain M, Pluchino N, Dallenbach P, Wenger JM, Savoldelli GL, Rehberg-Klug B, Dubuisson J. Fast-Track in Minimally Invasive Gynecology: A Randomized Trial Comparing Costs and Clinical Outcomes. Front Surg. 2021 Nov 11;8:773653. doi: 10.3389/fsurg.2021.773653. eCollection 2021. PMID 34859043

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT04839263/Prot_SAP_000.pdf